CLINICAL TRIAL: NCT04084951
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Dose Expansion Study of SQZ-PBMC-HPV as Monotherapy and in Combination With Atezolizumab or Other Immune Checkpoint Inhibitors in HLA-A*02+ Patients With HPV16+ Recurrent, Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of SQZ-PBMC-HPV in Patients With HPV16+ Recurrent, Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SQZ Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SQZ-PBMC-HPV-101
Record Dates: First submitted 2019-09-01; First posted 2019-09-10 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Adult Solid Tumor
Keywords: recurrent cancer; metastatic; locally advanced; cancer; cervical; head and neck; anal; penile; SQZ-PBMC-HPV; atezolizumab; HPV16; APC; cell therapy; ipilimumab; nivolumab; checkpoint inhibitors; immunotherapy; solid tumor; HLA-A*02; therapeutic vaccine; advanced solid tumor; rectal; vulvar; vaginal; PBMC; human papillomavirus strain 16; peripheral blood mononuclear cells; antigen presenting cells
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Neoplasms | interventions — atezolizumab; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Monotherapy Dose Escalation Phase (Experimental): In Part 1, SQZ-PBMC-HPV as a monotherapy is administered on Day 1 of every 3 week cycles for up to a year. In Cohort 3 (double-priming), SQZ-PBMC-HPV is also administered on Day 2 of Cycle 1. There are at least 3 groups ("Cohorts") in this Phase as follows:
  * Cohort 1: specified dose SQZ-PBMC-HPV
  * Cohort 2: specified dose SQZ-PBMC-HPV
  * Cohort 3: specified dose SQZ-PBMC-HPV double-priming
  Interventions: Biological: SQZ-PBMC-HPV
- Part 2 Combination Safety Phase (Experimental): In Part 2, SQZ-PBMC-HPV in combination with immune checkpoint inhibitors (1) atezolizumab, (2) ipilimumab, (3) nivolumab, or (4) nivolumab and ipilimumab, is administered every 3 weeks for up to a year except atezolizumab may be given up to 2 years; and ipilimumab will be administered four times (in a timeframe less than a year) if safety allows. There are 4 groups ("Cohorts") in this Phase as follows:
  * Cohort 4: SQZ-PBMC-HPV RP2D (Recommended Phase 2 Dose) plus atezolizumab
  * Cohort 5: SQZ-PBMC-HPV RP2D plus ipilimumab
  * Cohort 6: SQZ-PBMC-HPV RP2D plus nivolumab
  * Cohort 7: SQZ-PBMC-HPV RP2D plus nivolumab and ipilimumab
  Interventions: Biological: SQZ-PBMC-HPV; Drug: Atezolizumab; Drug: Ipilimumab; Drug: Nivolumab
- Part 3 Monotherapy Dose Expansion Phase (Experimental): In Part 3, SQZ-PBMC-HPV is administered at the RP2D to patients enrolled in HPV16+ cancer-type specific cohorts. There are 4 groups ("Cohorts") in this Phase as follows:
  * Cohort 8: SQZ-PBMC-HPV RP2D in HPV16+ head and neck cancer patients
  * Cohort 9: SQZ-PBMC-HPV RP2D in HPV16+ cervical cancer patients
  * Cohort 10: SQZ-PBMC-HPV RP2D in HPV16+ anal cancer patients
  * Cohort 11: SQZ-PBMC-HPV RP2D in other HPV16+ cancer patients
  Interventions: Biological: SQZ-PBMC-HPV

INTERVENTIONS:
Biological: SQZ-PBMC-HPV — antigen presenting cell therapy; therapeutic vaccine consisting of peripheral blood mononuclear cells (PBMCs) manufactured with immunogenic epitopes of HPV16
Drug: Atezolizumab — programmed cell death ligand 1 (PD-L1) blocking antibody
  Arms: Part 2 Combination Safety Phase
Drug: Ipilimumab — cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) blocking antibody
  Arms: Part 2 Combination Safety Phase
Drug: Nivolumab — programmed cell death 1 (PD-1) blocking antibody
  Arms: Part 2 Combination Safety Phase

SUMMARY:
This is a Phase 1 open-label, multicenter study of the safety and tolerability, immunogenic effects, antitumor activity, and pharmacodynamics of SQZ-PBMC-HPV as monotherapy and in combination with atezolizumab or other immune checkpoint inhibitors in HLA-A*02+ patients with recurrent, locally advanced or metastatic human papillomavirus strain 16 positive (HPV16+) solid tumors. The study includes patients with anal, rectal, cervical, head and neck, penile, vulvar, or vaginal cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients ≥18 years of age who are HLA-A*02+ (performed during screening locally or centrally, or based on documented historic test results)
* Histologically confirmed incurable or metastatic solid tumors that are HPV16+ (performed during screening locally or centrally, or based on documented historic test results)
* Cancer must have progressed after at least 1 available standard therapy for incurable disease, or the patient is intolerant to or refuses standard therapy(ies) or has a tumor for which no standard therapy(ies) exist
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1
* At least 1 measurable lesion according to RECIST 1.1
* Must have a lesion that can be biopsied with acceptable clinical risk and agree to have a fresh biopsy at Baseline and on Cycle 2 Day 8 (+/- 3 days)
* Patients must agree to venous access for the leukapheresis and be willing to have a central line inserted if venous access is an issue
* Adequate organ function and bone marrow reserve performed within 14 days prior to the leukapheresis

Exclusion Criteria:

* Treatment with anticancer therapy, including investigational therapy, within 2 weeks prior to leukapheresis. For prior therapies with a half-life longer than 3 days, discontinuation of the therapy must have occurred at least 28 days prior to leukapheresis
* Systemic treatment with either corticosteroids (>10 mg of prednisone or the equivalent per day) or other immunosuppressive medications within 14 days prior to leukapheresis
* Patients treated with non-corticosteroid based immunosuppressive agents within the last 6 months may not be eligible and should be discussed with the Sponsor
* Patients with active, known, or suspected autoimmune disease may not be eligible and should be discussed with the Sponsor
* Patients with >Grade 1 AEs related to previous treatment with anticancer or investigational therapy that do not resolve at least 2 weeks prior to leukapheresis, except neuropathy, ototoxicity, mucositis, fatigue, alopecia, or endocrine disorders managed with hormone replacement
* Known active hepatitis B or hepatitis C, or active mycobacterium tuberculosis infection
* History of any Grade 3 immune-related AE (irAE) from prior immunotherapy
* Has known active central nervous system metastases
* History of interstitial lung disease requiring steroids
* Major surgery within 2 weeks of leukapheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (TEAEs; all, related, serious, and of special interest) as assessed by CTCAE version 5.0 | Through 6 weeks after the patient's last dose of investigational product
  For SQZ-PBMC-HPV as a single agent (Part 1 and Part 3) and in combination with immune checkpoint inhibitors (Part 2)
Number of participants with dose-limiting toxicity (DLT) | Up to 1 year after LPFV
  For SQZ-PBMC-HPV as a single agent (Part 1 and Part 3) and in combination with immune checkpoint inhibitors (Part 2)
Objective response rate (ORR) [Part 3] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of complete response [CR] and/or partial response [PR] as defined by RECIST v1.1 criteria. For SQZ-PBMC-HPV as a single agent (Part 3 only)
Best overall response (BoR) [Part 3] | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product]
  Evaluation of the BoR defined as CR, PR, Stable Disease [SD], Progressive Disease [PD] or Not Evaluable [NE] as defined by RECIST v1.1 criteria. For SQZ-PBMC-HPV as a single agent (Part 3 only)
Progression-free survival (PFS) [Part 3] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Defined as the time from first dose of study treatment to first overall response of PD by RECIST v 1.1 or to death by any cause. This will be censored at the last RECIST v1.1 assessment if PD/death is not observed. For SQZ-PBMC-HPV as a single agent (Part 3 only)
Duration of Response (DoR) [Part 3] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Defined as the time from overall response of CR or PR to first overall response of PD by RECIST v1.1 or to death by any cause. This is defined only for patients who have a CR or PR and will be censored at the last RECIST v1.1 assessment if PD/Death is not observed. For SQZ-PBMC-HPV as a single agent (Part 3 only)
Disease-control rate (DCR) [Part 3] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of CR or PR or SD as defined by RECIST v1.1 criteria. For SQZ-PBMC-HPV as a single agent (Part 3 only)
Overall survival (OS) [Part 3] | Through study completion, up to 2 years
  Defined as the time from first dose of study treatment to death by any cause. This will be censored at the last date patient is known to be alive if death is not observed. For SQZ-PBMC-HPV as a single agent (Part 3 only)

SECONDARY OUTCOMES:
Objective response rate (ORR) [Part 1 and 2] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of complete response [CR] and/or partial response [PR] as defined by RECIST v1.1 criteria. For SQZ-PBMC-HPV as a single agent (Part 1) and in combination with immune checkpoint inhibitors (Part 2)
Best overall response (BoR) [Part 1 and 2] | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product]
  Evaluation of the BoR defined as CR, PR, Stable Disease [SD], Progressive Disease [PD] or Not Evaluable [NE] as defined by RECIST v1.1 criteria. For SQZ-PBMC-HPV as a single agent (Part 1) and in combination with immune checkpoint inhibitors (Part 2)
Progression-free survival (PFS) [Part 1 and 2] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Defined as the time from first dose of study treatment to first overall response of PD by RECIST v 1.1 or to death by any cause. This will be censored at the last RECIST v1.1 assessment if PD/death is not observed. For SQZ-PBMC-HPV as a single agent (Part 1) and in combination with immune checkpoint inhibitors (Part 2)
Duration of Response (DoR) [Part 1 and 2] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Defined as the time from overall response of CR or PR to first overall response of PD by RECIST v1.1 or to death by any cause. This is defined only for patients who have a CR or PR and will be censored at the last RECIST v1.1 assessment if PD/Death is not observed. For SQZ-PBMC-HPV as a single agent (Part 1) and in combination with immune checkpoint inhibitors (Part 2)
Disease-control rate (DCR) [Part 1 and 2] | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of CR or PR or SD as defined by RECIST v1.1 criteria. For SQZ-PBMC-HPV as a single agent (Part 1) and in combination with immune checkpoint inhibitors (Part 2)
Overall survival (OS) [Part 1 and 2] | Through study completion, up to 2 years
  For SQZ-PBMC-HPV as a single agent (Part 1) and in combination with immune checkpoint inhibitors (Part 2)
Amount of investigational product (IP) from individual patient blood collection [Part 1] | From leukapheresis through manufacture, a maximum of 28 days
  To determine manufacturing feasibility (Part 1 only)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - HonorHealth, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Anschutz Cancer Pavillion, Aurora, Colorado
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Masonic Cancer Center University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- University Hospital Cologne, Clinic I for Internal Medicine, Cologne, Germany